CLINICAL TRIAL: NCT00003262
Title: Prospective Non Randomized Study With Chemotherapy in Patients With Hodgkin's Disease and HIV Infection: "Stanford V Regimen" For "Low Risk" Patients, "EBVP Regimen" For "High Risk" Patients
Brief Title: Combination Chemotherapy in Treating Patients With Hodgkin's Disease and HIV Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066154; ITA-GICAT-POS5; EU-97022
Record Dates: First submitted 1999-11-01; First posted 2003-04-23 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2002-10

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; AIDS-related peripheral/systemic lymphoma; HIV-associated Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Filgrastim; Doxorubicin; Epirubicin; Etoposide; Mechlorethamine; Prednisone; Vinblastine; Vincristine

INTERVENTIONS:
Biological: bleomycin sulfate
Biological: filgrastim
Drug: Stanford V regimen
Drug: doxorubicin hydrochloride
Drug: epirubicin hydrochloride
Drug: etoposide
Drug: mechlorethamine hydrochloride
Drug: prednisone
Drug: vinblastine sulfate
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of two combination chemotherapy regimens in treating patients with Hodgkin's disease and HIV infection.

DETAILED DESCRIPTION:
OBJECTIVES:

* Investigate the effects on survival, life expectancy and quality, toxicity, and immunological status in low risk patients with Hodgkin's Disease and HIV infection treated with the Stanford V regimen and in high risk patients treated with epirubicin, bleomycin, vinblastine, and prednisone.

OUTLINE: Patients are stratified into 2 groups designated as low and high risk on the basis of ECOG performance status (0-2 vs 3-4), presence or absence of AIDS before the diagnosis of Hodgkin's Disease, and immune status (CD4+ cell count greater vs no greater than 100/mm^3).

* Low risk patients (those with no risk factors) receive the EBVP regimen, as follows:

  * Epirubicin intravenously on day 1
  * Bleomycin intramuscularly or intravenously on day 1
  * Vinblastine intravenously on day 1
  * Prednisone orally on days 1-5
  * Patients also receive daily injections of filgrastim (granulocyte colony-stimulating factor; G-CSF) on days 6-15. This schedule is repeated every 3 weeks for 6 courses.
* High risk patients (those with one or more risk factors) receive the Stanford V regimen, as follows:

  * Doxorubicin and vinblastine intravenously on days 1 and 15
  * Mechlorethamine intravenously on day 1
  * Vincristine and bleomycin intravenously on days 8 and 22
  * Etoposide intravenously on days 15 and 16
  * Prednisone orally daily
  * Patients also receive daily injections of G-CSF on days 3-7, 9-13, 17-21, and 23-26. This schedule is repeated every 28 days for 3 courses.

Patients are followed every 2 months the first year and then every 3 months thereafter.

PROJECTED ACCRUAL: 20-30 patients will initially be accrued in this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven Hodgkin's disease:

  * Clinical or pathologic stage II - IV
  * Stage I with bulky disease (tumor size greater than 10 cm) and B symptoms
* Confirmed HIV infection

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-4

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No severe cardiac disease

Pulmonary:

* No severe pulmonary disease

Other:

* No severe neurologic or metabolic disease
* No concurrent or prior second malignancy except:

  * Nonmelanomatous skin cancer
  * In situ cancer of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior therapy for Hodgkin's disease
* Concurrent triple-drug antiretroviral therapy (including one protease inhibitor) required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1997-05

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Tirelli, MD, Study Chair — Centro di Riferimento Oncologico - Aviano
Locations (1):
- Centro di Riferimento Oncologico - Aviano, Aviano, Italy

REFERENCES:
- [Background] Spina M, Gabarre J, Rossi G, Fasan M, Schiantarelli C, Nigra E, Mena M, Antinori A, Ammassari A, Talamini R, Vaccher E, di Gennaro G, Tirelli U. Stanford V regimen and concomitant HAART in 59 patients with Hodgkin disease and HIV infection. Blood. 2002 Sep 15;100(6):1984-8. doi: 10.1182/blood-2002-03-0989. PMID 12200356